CLINICAL TRIAL: NCT01901549
Title: Renal Denervation in Patients After Acute Coronary Syndrome
Acronym: ACSRD
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meshalkin Research Institute of Pathology of Circulation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AMIRD
Record Dates: First submitted 2013-07-08; First posted 2013-07-17 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Acute Coronary Syndrome; Arterial Hypertension
MeSH Terms: conditions — Acute Coronary Syndrome; Hypertension | interventions — Metoprolol; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PCI+Renal denervation (Active Comparator)
  Interventions: Procedure: Renal denervation; Drug: Metoprolol; Drug: Lisinopril
- PCI alone (Active Comparator)
  Interventions: Drug: Metoprolol; Drug: Lisinopril

INTERVENTIONS:
Procedure: Renal denervation — The treatment catheter is introduced into each renal artery and is applied discrete, radiofrequency ablations lasting up to 2 min each and of 8 watts or less to obtain up to six ablations separated both longitudinally and rotationally within each renal artery. During ablation, the catheter system monitored tip temperature and impedance, altering radiofrequency energy delivery in response to a predetermined algorithm. After the procedure the control arterial angiogram should be done.
  Arms: PCI+Renal denervation
Drug: Metoprolol — Beta-blockers. Optimal mediсal therapy will be assigned according to ACS and STE guidelines.
Drug: Lisinopril — ACE inhibitors. Optimal mediсal therapy will be assigned according to ACS and STE guidelines.

SUMMARY:
This study is aimed to evaluate the effect of renal denervation to decreasing blood pressure and left ventricle remodeling progression in patients after acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* acute Q negative myocardium infarction (during first 14 days)
* non stable angina
* significant stenosis
* BP > 140/90 torr. during more than 1 year

Exclusion Criteria:

* absence of arterial hypertension
* Thrombolysis during previous 24 hours
* indications for CABG

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2013-06; Primary Completion 2015-06 (Actual); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
cardiovascular death | 1 year
myocardium infarction | 1 year
stroke | 1 year
repeat revascularization | 1 year

SECONDARY OUTCOMES:
blood pressure changes | 1 year
CCS and NYHA | 1 year
heart rhythm disturbances | 1 year
intima-media index | 1 year
IVS thickness | 1 year
restenosis | 1 year
diastolic disfunction | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Evgeny Pokushalov, MD, PhD, Principal Investigator — State Research Institute of Circulation Pathology
Locations (1):
- State Research Institute of Circulation Pathology, Novosibirsk, Russia

REFERENCES:
- See also: State Research Institute of Circulation Pathology Official Site — http://meshalkin.ru